CLINICAL TRIAL: NCT04845594
Title: Randomized Efficacy Trial of MySmileBuddy, a Family-centered Behavioral Intervention to Reduce Early Childhood Caries
Brief Title: Efficacy Trial of MySmileBuddy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was halted prior to the start of enrollment due to the COVID-19 pandemic. The inability to conduct planned in-person intervention activities during the pandemic related to inherent risks of the virus necessitated withdrawal of the study.
Sponsor: Columbia University (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Carol Kunzel, Professor of Dental Community Health, Dental Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AAAR7549; 1U01DE026739-01A1 (NIH)
Record Dates: First submitted 2021-04-09; First posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Tooth Decay
Keywords: Oral hygiene; Decay; Decay Progression
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MySmileBuddy (Experimental): Children, aged 24-71 months of age, who have tooth decay will be enrolled, along with their caregiver, and will receive a family-focused intervention called MySmileBuddy.
  Interventions: Behavioral: MySmileBuddy (MSB)
- Control (No Intervention): Children, aged 24-71 months of age, who have tooth decay will be enrolled, along with their caregiver, and will not receive any intervention.

INTERVENTIONS:
Behavioral: MySmileBuddy (MSB) — The technology-based MSB program equips community health workers (CHWs) with an iPad-based app that facilitates assessment of a child's early childhood caries (ECC).
  Other Names: MSB
  Arms: MySmileBuddy

SUMMARY:
This study seeks to evaluate the best way to encourage a healthy diet and proper fluoride use in children at greatest risk for tooth decay. To do so, this study will evaluate whether or not a family focused intervention, MySmileBuddy, is able to reduce tooth decay progression in Hispanic preschoolers at high risk of this disease.

DETAILED DESCRIPTION:
Tooth decay in young children has traditionally been treated through surgical dental repair, an approach that does not address the oral hygiene and dietary behaviors that cause the disease. Professionals agree that behavioral strategies to prevent tooth decay are needed, but they have not been well studied in Hispanic children in the United States that have disproportionately high rates of this disease. Use of fluoridated toothpaste twice a day and consumption of a healthy diet can both prevent tooth decay and stop it from progressing.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 24 to 71 months of age, have a minimum of 12 teeth present, and have early childhood caries (ECC)
* Will reside in the New York City (NYC) metropolitan for the following 12 months
* Parents must be 18 years or older and must report having a cell phone with texting capabilities

Exclusion Criteria:

* Children with developmental delays or medical conditions that would impede oral dietary intake, at-home oral hygiene practices, or receipt of oral exams
* Children with parents who are under the age of 18 years of age, do not report having a mobile phone, do not plan to reside in the New York City (NYC) metropolitan area for the following 12 months
* Children of parents who do not provide consent to participate.

Ages: 24 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-12-02 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
Change in Number of Decayed, Missing, or Filled Teeth or Surfaces | 12 months post-randomization
  Early childhood caries status will be determined by visual examination, assisted by an examination light, mirror, and probe with caries experience defined by number of teeth (t) and surfaces (s) that either have decay (d), are missing due to decay (m), or have had a dental filling (f) due to a cavity.
Proportion of Participants with Early Childhood Caries Progression | 12 months post-randomization
  The number of decayed, missing, or filled teeth (dmft)/decayed filled surfaces (dfs) as a count variable will be measured to determine the proportion of participants who have a positive change in the number of dmft/dfs post-intervention.

SECONDARY OUTCOMES:
Change in Twice Daily Fluoridated Toothpaste Use | 12 months post-randomization
  Tooth brushing behaviors will be assess by asking parents a series of multiple choice and open-ended questions and direct observation of tooth brushing behavior measured using the Tooth Brushing Observation Scale (Collett, et al., 2016) at baseline (T1) and 12 months post-randomization (T2).
Change in Consumption of a Low Cariogenic Diet | 12 months post-randomization
  Cariogenic diet behaviors will be assessed by asking parents a series of multiple choice and open-ended questions using: (1) an age-appropriate modification of the University of Iowa's Diet Assessment of Caries Risk tool (Marshall, 2009); and (2) the MSB-developed modified 24-hour dietary recall widget.

CONTACTS AND LOCATIONS:
Overall Officials: Carol Kunzel, PhD, Principal Investigator — Columbia University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lumsden CL, Edelstein BL, Basch CE, Wolf RL, Koch PA, McKeague I, Leu CS, Andrews H. Protocol for a family-centered behavioral intervention to reduce early childhood caries: the MySmileBuddy program efficacy trial. BMC Oral Health. 2021 May 7;21(1):246. doi: 10.1186/s12903-021-01582-4. PMID 33962602